CLINICAL TRIAL: NCT00670683
Title: Safety and Efficacy of Insulin Detemir (Levemir® FlexPen®) in Patients With Diabetes Mellitus
Brief Title: Observational Study of Patients With Diabetes Using Levemir® FlexPen®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1914
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation

SUMMARY:
This study is conducted in Asia. This study is a prospective, open, uncontrolled, observational surveillance study with Levemir® FlexPen® conducted in Korea.

The aim of this observational study is to evaluate the short term and the long term safety and efficacy of Levemir® FlexPen®. The study is planned and conducted as per requirement from Korea Food and Drug Administration (KFDA).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus

Exclusion Criteria:

* Contra-indication based on local label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 797 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | for the duration of the trial

SECONDARY OUTCOMES:
Weight | for the duration of the trial
FBG (Fasting Blood Glucose) | for the duration of the trial
2hr-PPBG (2hr-Post Prandial Blood Glucose) | for the duration of the trial
HbA1c | for the duration of the trial
Adverse events | for the duration of the trial
Clinical laboratory abnormality | for the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Pusan, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com